CLINICAL TRIAL: NCT06873594
Title: Comparison of the Outcomes of Three Port and Four Port Laparoscopic Cholecystectomy in Patients Presenting to Tertiary Care Hospital: A Randomized Controlled Trial
Brief Title: Comparison of Three Ports and Four Ports Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical College, Peshawar (Other)
Responsible Party: Principal Investigator, Nisar Ahmed, Associate Professor Surgery, Khyber Medical College, Peshawar
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 163/DME/KMC
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cholelithiasis; Laparoscopic Cholecystectomy
Keywords: Three-port; Four-port; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- four-ports laparoscopic cholecystectomy (Active Comparator): in this arm, laparoscopic cholecystectomy will be done with three ports
  Interventions: Procedure: four-port laparoscopic cholecystectomy
- Three-port Laparoscopic cholecystectomy (Experimental): in this arm, laparoscopic cholecystectomy will be done with three ports
  Interventions: Procedure: three-ports laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: three-ports laparoscopic cholecystectomy — in this arm, laparoscopic cholecystectomy will be done with three ports
  Arms: Three-port Laparoscopic cholecystectomy
Procedure: four-port laparoscopic cholecystectomy — in this arm, laparoscopic cholecystectomy will be done with four ports
  Arms: four-ports laparoscopic cholecystectomy

SUMMARY:
Laparoscopic cholecystectomy is done traditionally with four ports. It has been observed that the same could be achieved using three ports. In this study we will study the outcomes of laparoscopic cholecystectomy done with both techniques.

DETAILED DESCRIPTION:
The gallbladder functions include the storage, concentration, and release of bile into the gut through synchronous contraction. Gallbladder disease is the predominant digestive disorder that may necessitate hospitalization. Gallbladder stones (cholelithiasis) are prevalent in adults, with a prevalence rate of 4.3% in India. The prevalence of gallstones, or cholelithiasis, in the adult population of ranges from 10% to 20% 1, 2.

In cases of chronic and acute calculus cholecystitis, complications arising from cholelithiasis, the preferred treatment is laparoscopic cholecystectomy, which offers diminished post-operative morbidity, lower complication rates, and expedited recovery, albeit with a slight elevation in conversion rates. Therefore, the preferred treatment for high-risk silent cholelithiasis, symptomatic cholelithiasis, persistent calculus cholelithiasis, as well as acute calculus cholelithiasis involves laparoscopic cholecystectomy 3, 4.

This method typically involves the creation of four small incisions in the abdomen, allowing for the introduction of a camera and surgical instruments to facilitate the dissection and removal of the gallbladder. The four-port technique offers several advantages, including improved visualization and maneuverability, which can be particularly beneficial in complex cases or when there are anatomical variations 5, 6. However, as surgical techniques evolve, the three-port laparoscopic cholecystectomy has emerged as a viable alternative, offering the potential for even less invasiveness and quicker recovery times. Proponents of the three-port technique argue that it results in less postoperative pain, reduced narcotic use, and faster recovery due to fewer incisions and reduced tissue trauma. It is observed that experienced surgeons have implemented numerous changes in laparoscopic cholecystectomy, including a reduction in port size. A cholecystectomy can be performed successfully without the utilization of four ports 7-9. A study compared the outcomes of three-port and four-port laparoscopic cholecystectomy i.e Mean pain score (2.19 + 1.06, and 2.91 + 1.20), Return to normal activity (4.9 + 0.85, and 5.8 + 1.95 ), and Post-operative hospital stay (1.19 + 0.06, and 1.44 + 0.17) 10.

As the three-port approach gains popularity due to its potential benefits, it comprehensive comparisons with the traditional four-port technique is essential to determine which technique is more clinically significant. As no such study is available on this subject locally, that is why the goal of this study is to compare the outcomes of three-port and four-port laparoscopic cholecystectomy at our health facility. Understanding the differences in overall patient outcomes can provide valuable insights for surgeons and patients alike, enabling informed decisions about the most appropriate surgical method based on individual patient conditions and the complexity of their gallbladder disease. This study will be helpful to bridge the knowledge gap regarding the efficacy and safety of both techniques, ultimately guiding clinical practice and enhancing patient care in laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cholelithiasis, scheduled for elective laparoscopic cholecystectomy
* both genders

Exclusion Criteria:

* conversion to open cholecystectomy
* patients requiring other bail-out procedures
* lactating and pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | 48 hours
  Mean pain score measured with a 0 to 10 scale visual analogue scale
Operative Time | same day of surgery
  Number of minutes of operative time

SECONDARY OUTCOMES:
Return to normal activity | 2 weeks
  Measured in number of days
hospital stay | 2 weeks
  post operative hospital stay measured in days

IPD SHARING:
Plan to Share IPD: Yes
Patients demographics, operative data and outcome data
Supporting Information: Study Protocol, SAP
Time Frame: 1 april 2025